CLINICAL TRIAL: NCT00250497
Title: New Moves: Obesity Prevention Among Adolescent Girls
Brief Title: New Moves - Obesity Prevention Among Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0309S51763; R01DK063107 (NIH)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Obesity
Keywords: Adolescent; Girls; Physical Activity; Exercise; Diet; Body image
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New Moves Intervention Group (Experimental): The New Moves intervention is an all girls physical education class that provides a supportive environment for girls. Girls participate in noncompetitive physical activities. They also receive lessons on nutrition and social support. After the class is over, girls continue to receive intervention messages through weekly lunch meetings. Girls meet individually with a personal coach.
  Interventions: Behavioral: New Moves
- control group (No Intervention): Girls in the control group participated in an all-girls physical education class but did not receive additional components offered in the intervention such as individual coaching.

INTERVENTIONS:
Behavioral: New Moves — The New Moves intervention is an all girls physical education class that provides a supportive environment for girls. Girls participate in noncompetitive physical activities. They also receive lessons on nutrition and social support. After the class is over, girls continue to receive intervention messages through weekly lunch meetings. Girls meet individually with a personal coach.
  Arms: New Moves Intervention Group

SUMMARY:
The New Moves study will evaluate the impact of a school based program for inactive high school girls who are overweight or at risk for being overweight due to low levels of physical activity. The primary study hypothesis is that girls in the intervention schools will significantly decrease their percent body fat as compared to girls in the control schools. Secondary research hypotheses include that girls in the intervention condition will significantly increase their physical activity levels and improve the quality of their dietary intake.

DETAILED DESCRIPTION:
The purpose of the New Moves study is to evaluate the effectiveness of a school-based all girls alternative to regular physical education class for inactive high school girls. New Moves uses a large-scale community randomized controlled study involving girls from six intervention schools and six control schools. The New Moves class includes physical activity, nutritional guidance, and social support within a supportive, non-competitive environment. In addition the program includes individual counseling sessions.

The primary research hypothesis is that girls in the intervention condition will significantly decrease their percent body fat as compared to girls in the control condition. Secondary research hypothesis to be tested are that girls in the intervention condition will significantly increase their level of physical activity and improve the quality of their dietary intake as compared to girls in the control condition. In addition a range of socioenvironmental, personal, and behavioral variables will be compared across conditions.

ELIGIBILITY:
Inclusion Criteria:

* High school girls
* Low levels of physical activity - defined as being in precontemplation, contemplation, or preparation stages of change for physical activity with activity levels at, or below, 30 minutes per day/three days per week outside of school physical education class
* Priority will be given to girls with a body mass index (BMI) greater than or equal to the 75th percentile for age and gender

Exclusion Criteria:

* BMI less than the 25th percentile for age and gender

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 356 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Neumark-Sztainer, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Division of Epidemiology and Community Health, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Neumark-Sztainer D, Flattum CF, Story M, Feldman S, Petrich CA. Dietary approaches to healthy weight management for adolescents: the New Moves model. Adolesc Med State Art Rev. 2008 Dec;19(3):421-30, viii. PMID 19227384
- [Result] Flattum C, Friend S, Neumark-Sztainer D, Story M. Motivational interviewing as a component of a school-based obesity prevention program for adolescent girls. J Am Diet Assoc. 2009 Jan;109(1):91-4. doi: 10.1016/j.jada.2008.10.003. PMID 19103327
- [Result] Neumark-Sztainer D, Bauer KW, Friend S, Hannan PJ, Story M, Berge JM. Family weight talk and dieting: how much do they matter for body dissatisfaction and disordered eating behaviors in adolescent girls? J Adolesc Health. 2010 Sep;47(3):270-6. doi: 10.1016/j.jadohealth.2010.02.001. Epub 2010 Apr 21. PMID 20708566
- [Result] Neumark-Sztainer DR, Friend SE, Flattum CF, Hannan PJ, Story MT, Bauer KW, Feldman SB, Petrich CA. New moves-preventing weight-related problems in adolescent girls a group-randomized study. Am J Prev Med. 2010 Nov;39(5):421-32. doi: 10.1016/j.amepre.2010.07.017. PMID 20965379
- [Result] Bauer KW, Neumark-Sztainer D, Fulkerson JA, Hannan PJ, Story M. Familial correlates of adolescent girls' physical activity, television use, dietary intake, weight, and body composition. Int J Behav Nutr Phys Act. 2011 Mar 31;8:25. doi: 10.1186/1479-5868-8-25. PMID 21453516
- [Result] Bauer KW, Neumark-Sztainer D, Fulkerson JA, Story M. Adolescent girls' weight-related family environments, Minnesota. Prev Chronic Dis. 2011 May;8(3):A68. Epub 2011 Apr 15. PMID 21477508
- [Result] Bauer KW, Neumark-Sztainer D, Hannan PJ, Fulkerson JA, Story M. Relationships between the family environment and school-based obesity prevention efforts: can school programs help adolescents who are most in need? Health Educ Res. 2011 Aug;26(4):675-88. doi: 10.1093/her/cyr027. Epub 2011 May 2. PMID 21536714
- [Result] Flattum C, Friend S, Story M, Neumark-Sztainer D. Evaluation of an individualized counseling approach as part of a multicomponent school-based program to prevent weight-related problems among adolescent girls. J Am Diet Assoc. 2011 Aug;111(8):1218-23. doi: 10.1016/j.jada.2011.05.008. PMID 21802570
- [Result] Meyer KA, Demerath EW, Friend S, Hannan PJ, Neumark-Sztainer D. Body fat is differentially related to body mass index in U.S.-born African-American and East African immigrant girls. Am J Hum Biol. 2011 Sep-Oct;23(5):720-3. doi: 10.1002/ajhb.21201. Epub 2011 Jul 25. PMID 21793092
- [Result] Meyer KA, Friend S, Hannan PJ, Himes JH, Demerath EW, Neumark-Sztainer D. Ethnic variation in body composition assessment in a sample of adolescent girls. Int J Pediatr Obes. 2011 Oct;6(5-6):481-90. doi: 10.3109/17477166.2011.596841. Epub 2011 Jul 12. PMID 21749194
- [Result] Bauer KW, Friend S, Graham DJ, Neumark-Sztainer D. Beyond Screen Time: Assessing Recreational Sedentary Behavior among Adolescent Girls. J Obes. 2012;2012:183194. doi: 10.1155/2012/183194. Epub 2011 Oct 12. PMID 22013514
- [Result] Friend S, Bauer KW, Madden TC, Neumark-Sztainer D. Self-weighing among adolescents: associations with body mass index, body satisfaction, weight control behaviors, and binge eating. J Acad Nutr Diet. 2012 Jan;112(1):99-103. doi: 10.1016/j.jada.2011.08.036. Epub 2011 Nov 4. PMID 22717180
- [Result] Friend S, Flattum CF, Simpson D, Nederhoff DM, Neumark-Sztainer D. The researchers have left the building: what contributes to sustaining school-based interventions following the conclusion of formal research support? J Sch Health. 2014 May;84(5):326-33. doi: 10.1111/josh.12149. PMID 24707927
- [Result] Graham DJ, Bauer KW, Friend S, Barr-Anderson DJ, Nuemark-Sztainer D. Personal, behavioral, and socio-environmental correlates of physical activity among adolescent girls: cross-sectional and longitudinal associations. J Phys Act Health. 2014 Jan;11(1):51-61. doi: 10.1123/jpah.2011-0239. Epub 2012 Dec 17. PMID 23250194

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: New Moves Intervention
- Control Group: All Girls PE Control group
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 182 | 174
Completed | 177 | 159
Not Completed | 5 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 182 | 174 | 356
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 174 | 165 | 339
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.13) | 15.8 (1.22) | 15.8 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 174 | 356
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 182 | 174 | 356

OUTCOME MEASURES:

1. Primary Outcome: Percent Body Fat
Description: Measured with DEX-A at baseline and 1 year follow-up
Time Frame: Baseline and One year
Measure: Mean (Standard Deviation); unit: % body fat (DXA)
Groups:
- Intervention Group: New Moves Intervention Group
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 177 | 159
% body fat (DXA) | 37.2 (9.55) | 37.7 (8.84)

2. Secondary Outcome: Level of Physical Activity
Description: The 3DPAR assessed the sedentary behaviors and physical activities that study participants engaged in during each half hour time block between 6 AM and midnight on the three days previous to the day of data collection. In order to complete the 3DPAR, participants were provided with a list of 65 common sedentary behaviors and physical activities and were asked to select the activity that they participated in for the majority of every 30-minute block. The number of blocks of physical activity were summed for each day and then averaged over the 3 days. Outcomes was the average # of 30 minute blocks of physical activity.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: average number of 30-minute blocks/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 177 | 159
average number of 30-minute blocks/day | 4.92 (3.52) | 3.72 (3.65)

3. Secondary Outcome: Fruits and Vegetables
Time Frame: One year
Measure: Mean (Standard Deviation); unit: Servings/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 177 | 159
Servings/day | 2.06 (2.18) | 1.82 (1.76)

4. Secondary Outcome: Sedentary Activity
Description: The 3DPAR assessed the sedentary behaviors and physical activities that study participants engaged in during each half hour time block between 6 AM and midnight on the three days previous to the day of data collection. In order to complete the 3DPAR, participants were provided with a list of 65 common sedentary behaviors and physical activities and were asked to select the activity that they participated in for the majority of every 30-minute block. The number of blocks of sedentary activity were summed for each day and then averaged over the 3 days. Outcomes was the average # of 30 minute blocks of sedentary activity per day
Time Frame: One Year
Measure: Mean (Standard Deviation); unit: average number of 30-minute blocks/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 177 | 159
average number of 30-minute blocks/day | 31.0 (3.82) | 32.3 (3.89)

5. Secondary Outcome: Unhealthy Weight Control Behaviors
Description: Ten questions assessing use of unhealthy weight control behaviors in the past month (yes/no). Behavior categories included fasted, ate very little, took diet pills, made myself vomit, used laxatives, used diuretics, used food substitutes, skipped meals, smoked more cigarettes, and went on a diet. If a respondent reported doing any of these behaviors, they were classified as having used unhealthy weight control behaviors.
Time Frame: One Year
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 177 | 159
percentage of participants | 49.5 | 63.3

6. Secondary Outcome: Body Satisfaction
Description: Ten questions assessing satisfaction with weight, height, and specific parts of the body; six Likert response categories.Body Satisfaction Scale Range=10-60 with higher values indicating increased body satisfaction.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 177 | 159
units on a scale | 40.7 (12.8) | 36.6 (12.4)

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/174
Other Adverse Events (participants affected / at risk) | 0/182 | 0/174

LIMITATIONS AND CAVEATS:
Control group also had all-girls PE. Some girls missing body composition data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes